CLINICAL TRIAL: NCT00537615
Title: A Phase 1 Open-Label Single-Radiolabeled Dose Study To Investigate The Absorption, Metabolism And Excretion Of [14C] PD 0332334 In Six Healthy Male Volunteers
Brief Title: An Open-label Study to Investigate the Absorption, Metabolism and Excretion of Radiolabeled PD 0332334 in Six Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A5361010
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — imagabalin

INTERVENTIONS:
Drug: PD 0332334
  Other Names: imagabalin

SUMMARY:
The purpose of this study is to investigate the absorption, metabolism and excretion of [14C] PD 0332334 to characterize plasma, fecal and urinary radioactivity and identify any metabolites of [14C] PD 0332334.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Healthy male subjects between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
2. Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.
4. Subjects who are willing and able to comply with scheduled confinement period, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the trial:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, orallergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Subjects enrolled in a previous radionucleotide study or who have received radiotherapy within 12 months prior to screening or such that total radioactivity would exceed acceptable dosimetry.
3. Subjects whose occupation requires exposure to radiation or monitoring of radiation exposure.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Radioactivity parameters in plasma and whole blood - Cmax , Tmax , AUCinf, AUClast, t1/2, CL/F and V/F.
Total 14C data in blood, urine and feces
Ratio of radioactivity in red blood cells to plasma (RBC/plasma)
Cumulative recovery of radioactivity in urine and feces
Identification of metabolites in feces, plasma and urine if possible
Plasma, urine and fecal PD 0332334 pharmacokinetic parameters - Cmax, Tmax, AUClast, AUCinf, t1/2, CL/F, V/F, CLR, Ae24 and Ae24(%)

SECONDARY OUTCOMES:
Pharmacokinetic analysis of metabolites if detectable

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361010&StudyName=An%20open-label%20study%20to%20investigate%20the%20absorption%2C%20metabolism%20and%20excretion%20of%20radiolabeled%20PD%200332334%20in%20six%20healthy%20male%20volunteers